CLINICAL TRIAL: NCT07158840
Title: A Single Arm, Multi-center, Phase II Study of AK112 in Non-squamous Non-small Cell Lung Cancer (NSCLC) Patients With Actionable Genomic Alterations (AGA) Who Have Failed to Previous Tyrosine Kinase Inhibitor (TKI) Treatment
Brief Title: AK112 in Non-squamous Non-small Cell Lung Cancer (NSCLC)Patients With Actionable Genomic Alterations (AGA) Who Have Failed to Previous Tyrosine Kinase Inhibitor (TKI) Treatment
Acronym: AGA TKI NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-215
Record Dates: First submitted 2025-08-14; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — AK112 Monotherapy

SUMMARY:
AK112 in non-squamous non-small cell lung cancer patients with actionable genomic alterations (AGA) who have failed to previous tyrosine kinase inhibitor (TKI) treatment

ELIGIBILITY:
Inclusion Criteria:

1. Signed the Informed Consent Form (ICF) voluntarily。
2. Participants must be aged between 18 and 75 years (inclusive), regardless of gender.
3. ECOG performance status of 0 or 1.
4. With a life expectancy of ≥3 months.
5. Histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) or metastatic (stage IV) non-squamous NSCLC.
6. Prior to enrollment, participants must have at least one actionable genomic alteration (AGA) confirmed by tumor histology, cytology, or blood-based testing, including: EGFR, ALK, ROS1, NTRK, RET, BRAF and MET. Participants must provide a prior AGA test report; otherwise, AGA testing must be performed at the study site or at a site-designated laboratory before enrollment.
7. Previous treatment failure with an AGA-targeted TKI.
8. At least one measurable extracranial lesion as defined by RECIST v1.1.
9. Adequate organ function confirmed.

Exclusion Criteria:

1. Histological or cytological pathology confirming the presence of a small-cell carcinoma component or a predominant squamous cell carcinoma component.
2. AGA test report showing the presence of a common EGFR sensitizing mutation.
3. Prior receipt of immunotherapy.
4. Prior receipt of any systemic anti-tumor therapy for advanced-stage (IIIB-IV) NSCLC other than AGA-targeted TKIs.
5. Concurrent participation in another clinical study, unless it is a non-interventional study or the follow-up phase of an interventional study.
6. Receipt of AGA-targeted TKI therapy within 2 weeks prior to the first dose; receipt of non-specific immunomodulatory therapy within 2 weeks prior to the first dose.
7. Imaging during the screening period shows tumor encasement of major blood vessels or significant necrosis/cavitation, and the investigator determines that study participation would pose a bleeding risk.
8. Imaging during the screening period shows tumor invasion of surrounding vital organs or blood vessels.
9. Central nervous system metastases: participants assessed by the investigator as not requiring local treatment may be eligible; leptomeningeal metastases are not eligible.
10. History of malignancy other than NSCLC within 3 years prior to the first dose; participants with other malignancies that have been cured by local treatment are allowed.
11. Active autoimmune disease requiring systemic therapy within 2 years prior to the first dose.
12. History of major medical conditions within 1 year prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Overall response (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by investigator | up to 2 years
  Proportion of subjects who have a complete or partial response as assessed according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  From date of enrollment until the date of death from any cause
Progression-free survival (PFS) | up to 2 years
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first
Duration of response (DoR) | up to 2 years
  Duration of response (DoR), which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | up to 2 years
  Disease control rate (DCR), which is defined as the proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD), based on RECIST v1.1
Time to response (TTR) | up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
Percentage of participants with adverse event (AE) | From the subject signs the Informed Consent Form to 30 days (AE) and 90 days (Serious AE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first,up to 2 years
  The percentage of participants experiencing an adverse event (AE) and the severity of AEs will be assessed
Observed concentrations of AK112 | From date of enrollment until the end of treatment, assessed up to 2 years
  The endpoints for assessment of Pharmacokinetics (PK) of AK112 include serum concentrations of AK112 at different timepoints after AK112 administration
Number of participants who develop detectable anti-drug antibodies (ADAs) | From first dose of AK112 through 90 days after last dose of AK112,up to 2 years
  The immunogenicity of AK112 will be assessed by summarizing the number of participants who develop detectable antidrug antibodies (ADAs)
Number of participants with programmed cell death ligand 1 (PD-L1) expression positive who achieve CR/PR | From date of enrollment until the end of treatment, assessed up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, China